CLINICAL TRIAL: NCT04802330
Title: PREVALENCE OF FEMALE GENITAL MUTILATION IN BENI SUEF LOCALITIES
Brief Title: PREVALENCE OF FEMALE GENITAL MUTILATION IN BENI-SUEF LOCALITIES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Professor in Obstetrics and Gynecology Department, Beni-Suef University
Other Study IDs: Beni-Suef 21
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Female Genital Mutilation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female genital mutilation: Assessment of FGM prevalence in Beni Suef localities and its impact on studied women.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Assessment of causes of FGM Beni Suef localities. 3. Explore the relationship between some of the social and demographic variables such as age, education, place of residence, marital status, religion and economic level and practice of FGM.

SUMMARY:
Female genital mutilation /cutting (FGMC) includes all procedures that involve partial or total removal of the external female genitalia, or another injury to the female genital organs for non-medical reasons". It constitutes an extreme form of discrimination against women due to the health consequences, pain, and risks involved. Regardless of its prevalence, the physical and psychological complications of FGM in Egypt were shown to be enormous. These complications are usually categorized into primary or acute complications and secondary or long-term complications. The primary complications include pain, bleeding, and psychiatric trauma while the secondary complications include several emotional, menstrual, and sexual disorders

DETAILED DESCRIPTION:
Despite being internationally recognized as a human rights violation of girls and women, FGM has been performed on at least 200 million girls and women in 31 countries. According to the 2015 Egypt Health Issues Survey (EHIS), 87% of all women aged 15-49 years in Egypt had undergone FGM. Social norms, religion, ensuring premarital virginity and marital fidelity, increasing marriageability, and cultural ideals of femininity and modesty were among the most commonly cited reasons for performing FGM. A survey conducted among Egyptians aged 10-29 years in 2014 indicated that the reasons given for practicing FGM were customs and traditions (56.7%) and religion (35%).

FGM has many types ranging from excision of the prepuce with/out clitoris (Type I or Clitoridectomy) and excision of the clitoris and labia minora (Type II or Excision) to profound excision of the external genitalia with stitching and tightening the vaginal opening (Type III or Infibulation). Type IV describes pricking, piercing, scraping, and cauterization of the external genitalia without flesh removal. In societies with Muslim majorities, type I: is known as "Sunna Circumcision"; a religious term linking the practice to the commands of the Prophet of Islam or "Khifad" the Arabic synonym of "reduction"; a term claiming that the Prophet of Islam endorsed partial rather than complete excision of the external genitalia. In Egypt, types I and II are also called "Ta-hara"; the Arabic synonym of "purification" which points to the hygienic drive of the practice.

ELIGIBILITY:
Inclusion Criteria:

* Living in Beni Suef Governorate.

Exclusion Criteria:

* Women and men who complaining of any psychological problems

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consisted of all males and females who will be attended to the previously mentioned study setting at the time of data collection will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the impact of FGM | During 13 months
  The investigators will evaluate the consequences of female genital mutilation on participants of the study.
To estimate intention to practice FGM | During 13 months
  The participants will be given questions concerning intention to practice FGM in future. This section included questions regarding females' plans of mutilating their daughters in future, whether they were facing social pressure from family members or neighbors, whether they knew someone who intended to mutilate their daughters.

SECONDARY OUTCOMES:
To collect information about history of circumcision for the woman and her daughter. | During 13 months
  A questionnaire rituals of FGM and the decision-maker.

CONTACTS AND LOCATIONS:
Locations (1):
- Nesreen Abdel Fattah Abdallah Shehata, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdou, Marwa SM, Iman MH Wahdan, and Nessrin A. El-Nimr.
- [Background] Shell-Duncan B. The medicalization of female "circumcision": harm reduction or promotion of a dangerous practice? Soc Sci Med. 2001 Apr;52(7):1013-28. doi: 10.1016/s0277-9536(00)00208-2. PMID 11266046
- [Background] Tag-Eldin MA, Gadallah MA, Al-Tayeb MN, Abdel-Aty M, Mansour E, Sallem M. Prevalence of female genital cutting among Egyptian girls. Bull World Health Organ. 2008 Apr;86(4):269-74. doi: 10.2471/blt.07.042093. PMID 18438515